CLINICAL TRIAL: NCT00311090
Title: International, Multicenter, Randomized, Parallel Group, Double-blind Study, in Patients With Acute Symptomatic Deep Vein Thrombosis of the Lower Limbs, Demonstrating the Bioequipotency at Steady State of Equimolar Doses of SSR126517E (3.0 mg) Once a Week and SR34006 (2.5 mg) Once a Week, Documenting the Safety and Efficacy of Both Compounds During a 6-month Treatment, and Demonstrating the Neutralizing Effect of SSR29261 on the SSR126517E-induced Anti-Xa Activity
Brief Title: Bioequipotency Study of Idrabiotaparinux and Idraparinux in Patients With Deep Venous Thrombosis of the Lower Limbs
Acronym: EQUINOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC5945; 2005-005326-30 (EudraCT Number)
Record Dates: First submitted 2006-04-04; First posted 2006-04-05 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-02

CONDITIONS: Deep Venous Thrombosis
Keywords: Deep Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — idraparinux; Avidin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Idrabiotaparinux (Experimental): Idrabiotaparinux sodium , 3.0 mg, once-weekly for 6 months.
  In avidin sub-study, participants receive on Day 183, avidin 100 mg or placebo (for avidin) (4 hours after Idrabiotaparinux administration)
  Interventions: Drug: Idrabiotaparinux sodium; Drug: Avidin; Drug: Placebo (for Avidin)
- Idraparinux (Active Comparator): Idraparinux sodium, 2.5 mg, once-weekly for 6 months
  In avidin sub-study, participants receive on Day 183, placebo (for avidin) (4 hours after Idrabiotaparinux administration)
  Interventions: Drug: Idraparinux sodium; Drug: Placebo (for Avidin)

INTERVENTIONS:
Drug: Idrabiotaparinux sodium — 0.5 mL pre-filled syringe for 3.0 mg
  Subcutaneous injection
  Other Names: Biotinylated Idraparinux; SSR126517
  Arms: Idrabiotaparinux
Drug: Idraparinux sodium — 0.5 mL pre-filled syringe for 2.5 mg
  Subcutaneous injection
  Other Names: SR34006
  Arms: Idraparinux
Drug: Avidin — 100 mg in 10 mg/mL solution
  Intravenous infusion for 30 minutes
  Other Names: SSR29261
  Arms: Idrabiotaparinux
Drug: Placebo (for Avidin) — Avidin matching powder in 10 mg/mL solution
  Intravenous infusion for 30 minutes

SUMMARY:
The three purposes of this study are the following:

* To compare during a 6-month treatment the safety and effectiveness of idrabiotaparinux (SSR126517) with that of idraparinux (SR34006), taking into account new events of deep venous thrombosis (DVT) and pulmonary embolism (PE), and bleeding risk;
* To compare the activities of idrabiotaparinux and idraparinux directly in blood during and after a 6-month treatment;
* To check the ability of avidin (SSR29261) to reverse the blood thinning activity of idrabiotaparinux at the end of a 6-month treatment period.

DETAILED DESCRIPTION:
The study consists in a 6-month treatment period followed by an observational period of 3 to 6 months with a month 9 visit and a phone/contact visit at month 12.

All participants who complete the 6-month treatment period are re-randomized to either the idrabiotaparinux/idraparinux bioequipotency sub-study or the avidin neutralizing effect sub-study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed acute symptomatic DVT of the lower limbs

Exclusion Criteria:

* Severe concomitant diseases (e.g. renal failure, hepatic failure, uncontrolled hypertension)
* Active bleeding or high risk for bleeding.
* Pregnancy or childbearing potential without proper contraceptive measures.
* Breastfeeding
* Known allergy to idraparinux, SSR126517E, or egg proteins
* Indication of prolonged anticoagulation for other reason than DVT of the lower limbs
* Symptomatic pulmonary embolism (PE)
* Life expectancy < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Bioequipotency sub-study: idrabiotaparinux/idraparinux ratio for pharmacodynamic exposure parameters | Day 183
Avidin neutralizing effect substudy: decrease in anti-Xa activity between the start and end of the avidin infusion | Day 183 to Day 188

SECONDARY OUTCOMES:
Pharmacokinetic profile: idrabiotaparinux and idraparinux plasma concentrations | Days 15, 36, 57, 92 and 183
Safety: number of participants with clinically relevant bleedings and number of deaths as confirmed by a Central Independent Adjudication Committee (CIAC) | First 6 months
Efficacy: number of participants with symptomatic recurrent venous thromboembolism as confirmed by the CIAC | First 6 months

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (20):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Buenos Aires, Argentina
- Sanofi-Aventis, Macquarie Park, Australia
- Sanofi-Aventis, Vienna, Austria
- Sanofi-Aventis, Diegem, Belgium
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Prague, Czechia
- Sanofi-Aventis, Copenhagen, Denmark
- sanofi-aventis France, Paris, France
- sanofi-aventis Israel, Netanya, Israel
- Sanofi-aventis, Milan, Italy
- sanofi-aventis Mexico, México, Mexico
- sanofi-aventis, Netherlands, Gouda, Netherlands
- Sanofi-Aventis, New Zealand, New Zealand
- Sanofi-Aventis, Warsaw, Poland
- Sanofi-aventis, Moscow, Russia
- Sanofi-Aventis, Midrand, South Africa
- Sanofi-Aventis, Barcelona, Spain
- sanofi-aventis Turkey, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Equinox Investigators. Efficacy and safety of once weekly subcutaneous idrabiotaparinux in the treatment of patients with symptomatic deep venous thrombosis. J Thromb Haemost. 2011 Jan;9(1):92-9. doi: 10.1111/j.1538-7836.2010.04100.x. PMID 20946157
- [Derived] Trellu M, Fau JB, Cortez P, Cheng S, Paty I, Boelle E, Donat F, Sanderink GJ. Bioequipotency of idraparinux and idrabiotaparinux after once weekly dosing in healthy volunteers and patients treated for acute deep vein thrombosis. Br J Clin Pharmacol. 2013 May;75(5):1255-64. doi: 10.1111/bcp.12009. PMID 23078631
- [Derived] Paty I, Trellu M, Destors JM, Cortez P, Boelle E, Sanderink G. Reversibility of the anti-FXa activity of idrabiotaparinux (biotinylated idraparinux) by intravenous avidin infusion. J Thromb Haemost. 2010 Apr;8(4):722-9. doi: 10.1111/j.1538-7836.2010.03746.x. Epub 2010 Jan 17. PMID 20088937